CLINICAL TRIAL: NCT04085536
Title: Multicenter Prospective Longitudinal Study on the Efficacy of Exclusive Odontological and Medical Treatment in the Management of Chronic Dental Maxillary Sinusitis
Brief Title: Prospective Study on the Efficacy of Exclusive Odontological and Medical Treatment in Chronic Dental Maxillary Sinusitis
Acronym: DENTASINUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENTASINUS
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Chronic Maxillary Sinusitis
MeSH Terms: interventions — Dental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic maxillary sinusitis(for more than 12 weeks) (Other): Patients for whom chronic maxillary sinusitis will be diagnosed in the first ENT consultation, will then be seen in a stomatology consultation to determine whether or not a dental cause is objective.
  Interventions: Procedure: Dental and medical treatment

INTERVENTIONS:
Procedure: Dental and medical treatment — If the dental cause of sinusitis is objective, if necessary, dental treatment combined with medical treatment will be carried out.

SUMMARY:
The study will be offered to patients for whom chronic maxillary sinusitis will be diagnosed in the first ENT (ear, nose and throat) consultation. These patients will then be seen in a stomatology consultation to determine whether or not a dental cause is objective

DETAILED DESCRIPTION:
Chronic maxillary sinusitis is an inflammatory condition and/or infectious diseases of the maxillary sinus, which last longer than 12 weeks. Those whose the origin is dental, are well described, and yet under-diagnosed most of the time due to a lack of well-defined diagnostic criteria and literature. There is controversy in the various studies about their prevalence. Their management and in particular the therapeutic sequence, is not the subject of any recommendation and involves only a few clinical studies. Their consequences on the patient's general health and quality of life are important. The lack of knowledge about them often leads to diagnostic errors and therefore to a persistence of symptomatology. Moreover, their complications when they are not or incorrectly treated, although rare, can be dramatic (occulo-orbital or endo-cranial complications for example).

Preliminary work in the form of a retrospective study was carried out within of the Centre Hospitalier intercommunal de Créteil in 2015. In view of the results the investigators wanted to set up a clinical trial with the following objectives measure the prevalence of chronic maxillary sinusitis of dental origin and measure the effectiveness of exclusive dental and medical treatment, which could avoid surgical intervention under general anaesthesia, at the higher morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Signed Informed Consent
3. Patient with chronic maxillary sinusitis diagnosed by examination of the patient and ENT examination by naso-fibroscopy
4. Sinus imaging to confirm the diagnosis (facial mass scanner or cone beam CT)
5. Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

1. Fungal bullet sinusitis
2. Naso-sinus polyposis
3. atelectasic sinusitis
4. Systemic damage that may affect the maxillary sinuses (muciviscidosis, primary ciliary dyskinesia, vasculitis, granulomatosis, history of radiotherapy of the facial mass, pregnancy)
5. Long-term immunosuppressive treatment (chemo, anti-rejection)
6. Rhinosinusian tumor process
7. Fronto-ethmoidomaxillary sinusitis with risk of orbital or meningeal damage in the short to medium term.
8. Refusal of consent
9. Simultaneous participation in another intervention research
10. Patient under guardianship, curatorship or justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of therapeutic successes | 3 months after the end of dental care
  Disappearance of symptoms and absence of pus from the meatus observed at the 2nd consultation visit ENT control

SECONDARY OUTCOMES:
Number of dental origin | 3 months after the end of dental care
  Patients whose dental origin has been identified
Percentage of patients with preserved teeth | 3 months after the end of dental care
  Percentage of patients who received conservative treatment of the tooth versus non-conservative dental treatment
Percentage of each type of dental disease causing chronic maxillary sinusitis | 3 months after the end of dental care
  Measure the prevalence of the different dental diseases that cause sinusitis

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hopitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Groupe Hospitalier Intercommunal Le Raincy-Montfermeil, Montfermeil

IPD SHARING:
Plan to Share IPD: No